CLINICAL TRIAL: NCT00321685
Title: Phase II Study of Preoperative Radiation With Concurrent Capecitabine, Oxaliplatin and Bevacizumab Followed by Surgery and Postoperative 5-FU, Leucovorin, Oxaliplatin (FOLFOX) and Bevacizumab in Patients With Locally Advanced Rectal Cancer
Brief Title: Bevacizumab, Radiation Therapy, and Combination Chemotherapy in Treating Patients Who Are Undergoing Surgery for Locally Advanced Nonmetastatic Rectal Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NCI-2009-01081; NCI-2009-01081 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); CDR0000471148; ECOG-E3204; E3204 (Other: ECOG-ACRIN Cancer Research Group); E3204 (Other: CTEP); U10CA180820 (NIH); U10CA021115 (NIH)
Record Dates: First submitted 2006-05-02; First posted 2006-05-04 (Estimated); Results first posted 2015-05-12 (Estimated); Last update posted 2019-03-27 (Actual); Status verified 2019-03

CONDITIONS: Rectal Adenocarcinoma; Stage II Rectal Cancer AJCC v7; Stage III Rectal Cancer AJCC v7
MeSH Terms: conditions — Rectal Neoplasms | interventions — Bevacizumab; Immunoglobulin G; Disulfides; Capecitabine; Fluorouracil; dehydroftorafur; Leucovorin; Oxaliplatin; Radiotherapy; Radiation

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Treatment (bevacizumab and chemoradiotherapy) (Experimental): See Detailed Description
  Interventions: Biological: Bevacizumab; Drug: Capecitabine; Drug: Fluorouracil; Drug: Leucovorin Calcium; Drug: Oxaliplatin; Radiation: Radiation Therapy; Procedure: Therapeutic Conventional Surgery

INTERVENTIONS:
Biological: Bevacizumab — Given IV
  Other Names: Anti-VEGF; Anti-VEGF Humanized Monoclonal Antibody; Anti-VEGF rhuMAb; Avastin; Bevacizumab Biosimilar BEVZ92; Bevacizumab Biosimilar BI 695502; Bevacizumab Biosimilar CBT 124; Bevacizumab Biosimilar FKB238; Bevacizumab Biosimilar MIL60; Bevacizumab Biosimilar QL 1101; BEVACIZUMAB, LICENSE HOLDER UNSPECIFIED; Immunoglobulin G1 (Human-Mouse Monoclonal rhuMab-VEGF Gamma-Chain Anti-Human Vascular Endothelial Growth Factor), Disulfide With Human-Mouse Monoclonal rhuMab-VEGF Light Chain, Dimer; Recombinant Humanized Anti-VEGF Monoclonal Antibody; rhuMab-VEGF
Drug: Capecitabine — Given PO
  Other Names: Ro 09-1978/000; Xeloda
Drug: Fluorouracil — Given IV
  Other Names: 5-Fluoro-2,4(1H, 3H)-pyrimidinedione; 5-Fluorouracil; 5-Fluracil; 5-FU; AccuSite; Carac; Fluoro Uracil; Fluouracil; Flurablastin; Fluracedyl; Fluracil; Fluril; Fluroblastin; Ribofluor; Ro 2-9757; Ro-2-9757
Drug: Leucovorin Calcium — Given IV
  Other Names: Adinepar; Calcifolin; Calcium (6S)-Folinate; Calcium Folinate; Calcium Leucovorin; Calfolex; Calinat; Cehafolin; Citofolin; Citrec; citrovorum factor; Cromatonbic Folinico; Dalisol; Disintox; Divical; Ecofol; Emovis; Factor, Citrovorum; Flynoken A; Folaren; Folaxin; FOLI-cell; Foliben; Folidan; Folidar; Folinac; Folinate Calcium; folinic acid; Folinic Acid Calcium Salt Pentahydrate; Folinoral; Folinvit; Foliplus; Folix; Imo; Lederfolat; Lederfolin; Leucosar; leucovorin; Rescufolin; Rescuvolin; Tonofolin; Wellcovorin
Drug: Oxaliplatin — Given IV
  Other Names: 1-OHP; Ai Heng; Aiheng; Dacotin; Dacplat; Diaminocyclohexane Oxalatoplatinum; Eloxatin; Eloxatine; JM-83; Oxalatoplatin; Oxalatoplatinum; RP 54780; RP-54780; SR-96669
Radiation: Radiation Therapy — Undergo radiotherapy
  Other Names: Cancer Radiotherapy; Irradiate; Irradiated; irradiation; Radiation; Radiotherapeutics; RADIOTHERAPY; RT; Therapy, Radiation
Procedure: Therapeutic Conventional Surgery — Undergo surgical resection

SUMMARY:
This phase II trial studies how well giving bevacizumab, radiation therapy, and combination chemotherapy works in treating patients who are undergoing surgery for locally advanced nonmetastatic rectal cancer. Monoclonal antibodies, such as bevacizumab, can block tumor growth in different ways. Some find tumor cells and kill them or carry tumor-killing substances to them. Others interfere with the ability of tumor cells to grow and spread. Bevacizumab may also stop the growth of tumor cells by blocking blood flow to the tumor. Radiation therapy uses high-energy x-rays to kill tumor cells. Drugs, such as capecitabine, may make tumor cells more sensitive to radiation therapy. Drugs used in chemotherapy, such as capecitabine, oxaliplatin, fluorouracil, and leucovorin, work in different ways to stop the growth of tumor cells, either by killing the cells or by stopping them from dividing. Giving bevacizumab together with radiation therapy and combination chemotherapy before surgery may make the tumor smaller and reduce the amount of normal tissue that needs to be removed. Giving bevacizumab together with combination chemotherapy after surgery may kill any tumor cells that remain after surgery.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To evaluate the pathological complete response rate in patients with T3 and T4 rectal cancers when treated preoperatively with capecitabine, oxaliplatin, bevacizumab, and concurrent radiotherapy (XRT).

II. To evaluate the resection rate for T3 and T4 rectal cancers and the expected versus actual type of resection (abdominoperinal resection [APR] vs. low anterior resection [LAR] vs. LAR/coloanal anastomosis).

III. To make preliminary observations of patient survival and patterns of recurrence for this treatment combination.

IV. To gain additional experience regarding the toxicity and tolerability of this preoperative and postoperative regimen.

OUTLINE:

PREOPERATIVE CHEMORADIOTHERAPY: Patients undergo radiotherapy (total dose to the tumor bed was 5040 cGy) once daily (QD) 5 days a week and receive capecitabine 825 mg/m^2 orally (PO) twice daily (BID) 5 days a week for 5.5 weeks. Patients also receive oxaliplatin 50 mg/m^2 intravenously (IV) over 2 hours on days 1, 8, 15, 22, and 29 and bevacizumab 5 mg/kg IV over 30-90 minutes on days 1, 15, and 29 during radiotherapy.

SURGERY: Approximately 6-8 weeks after completion of chemoradiotherapy, patients undergo surgical resection. Patients whose tumors are not completely resected or who have metastatic disease discontinue protocol therapy.

POSTOPERATIVE CHEMOTHERAPY: Approximately 4-12 weeks after surgery, patients receive oxaliplatin IV over 2 hours, leucovorin calcium 400 mg/m^2 IV over 2 hours, and bevacizumab 5 mg/kg IV over 30-90 minutes on day 1. Patients also receive fluorouracil 2400 mg/m^2 IV continuously over 46 hours beginning on day 1. Treatment repeats every 2 weeks for 9 courses in the absence of disease progression or unacceptable toxicity. Patients then receive up to 3 additional courses of leucovorin calcium, fluorouracil, and bevacizumab.

After completion of study treatment, patients are followed up periodically for 10 years.

ELIGIBILITY:
Inclusion Criteria:

* Patients must have histologically confirmed, locally advanced, non-metastatic primary T3 or T4 adenocarcinoma of the rectum
* Patients must not have evidence of tumor outside of the pelvis including liver metastases, peritoneal seeding, or metastatic inguinal lymphadenopathy
* Patients must not have intra-operative radiotherapy (IORT) or brachytherapy treatment to the pelvis
* The distal border of the tumor must be at or below the peritoneal reflection, defined as within 12 centimeters of the anal verge by proctoscopic examination
* Transmural penetration of tumor through the muscularis propria must be demonstrated by either of the following: computed tomography (CT) scan plus endorectal ultrasound, or a magnetic resonance imaging (MRI); an endorectal coil or pelvic MRI is allowed
* For the patient to be eligible, the surgeon must prospectively define the tumor as either initially resectable or potentially resectable after pre-operative chemoradiation; clinically resectable tumors are defined as completely resectable with negative margins based on routine examination of the non-anesthetized patient; patients whose tumors are not resectable are not eligible; before pre-operative (op) treatment, the surgeon should estimate and record the type of resection anticipated: pelvic exenteration, posterior pelvic exenteration, APR, LAR, or LAR/coloanal anastomosis
* Patients with tumors that are clinically fixed, clinical stage T4N0-2, M0 are eligible if it is believed that their tumors are potentially resectable after chemoradiation; based on the following:

  * Clinically fixed tumors on rectal examination with tumor adherent to the pelvic sidewall or sacrum
  * Sciatica attributed to sacral root invasion with CT scan/MRI evidence of the lack of clear tissue plane will be considered evidence of fixation
  * Hydronephrosis on CT scan or intravenous pyelogram (IVP) or ureteric or bladder invasion as documented by cystoscopy and cytology or biopsy, or invasion into prostate
  * Vaginal or uterine involvement
* Patients must have Eastern Cooperative Oncology Group (ECOG) performance status 0-1
* A surgical evaluation must confirm patient's ability to tolerate the proposed surgical procedure
* Patients must have a caloric intake > 1500 kilocalories/day (d)
* Within 4 weeks prior to registration, the patient's absolute neutrophil count (ANC) level must be >= 1,500/mm^3
* Within 4 weeks prior to registration, the patients platelet level must be >= 100,000/mm^3
* Within 4 weeks prior to registration, serum creatinine must be < 1.5 X upper limit of normal (ULN); if serum creatinine > 1.5 x ULN, then creatinine clearance must be >= 50 mL/mm
* Within 4 weeks prior to registration, serum bilirubin must be =< 1.5 X ULN
* Within 4 weeks prior to registration, alkaline phosphatase (alk phos) must be < 2 x ULN
* Within 4 weeks prior to registration, serum glutamic oxaloacetic transaminase (SGOT) must be < 2 x ULN
* Carcinoembryonic antigen (CEA) must be determined prior to initiation of therapy
* Within 4 weeks prior to registration, urine protein/creatinine (UPC) ratio must be < 1; patients with a ratio of >= 1 must undergo a 24-hour urine collection which must be an adequate collection and must demonstrate < 1 gram (gm) of protein in order to participate
* Within 4 weeks prior to registration, albumin must be >= 2 gm/dl
* Absence of clinical evidence of high-grade (lumen diameter < 1 cm) large bowel obstruction, unless diverting colostomy has been performed
* Eligible patients of reproductive potential (both sexes) must agree to use an accepted and effective method of contraceptive during study therapy and for at least 6 months after the completion of bevacizumab
* Women must not be pregnant or breast-feeding; all females of childbearing potential must have a serum pregnancy test to rule out pregnancy within 2 weeks of registration
* Patients must have had no prior chemotherapy for rectal cancer or pelvic irradiation therapy
* Patients with prior malignancies, including pelvic cancer, are eligible if they have been disease free for > 5 years; patients with prior in situ carcinomas are eligible provided there was complete removal
* Patients must have no active inflammatory bowel disease or other serious medical illness or disease that might limit the patient's ability to receive protocol therapy
* Patients with a history of cerebrovascular accident (CVA)/transient ischemic attack (TIA) at any time, or myocardial infarction/unstable angina within 12 months of study entry are not eligible
* Patients with > grade 1 peripheral neuropathy are not eligible
* Patients must have urine protein/creatinine (UPC) ratio of < 1.0; patients with a UPC ratio >= 1.0 must undergo a 24-hour urine collection, which must be an adequate collection and must demonstrate < 1 gm of protein in order to participate
* Patients with a history of hypertension must measure < 150/90 mmHg and be on a stable regimen of anti-hypertensive therapy
* Patients with clinically significant peripheral vascular disease are not eligible
* Patients must not have any of the following:

  * Unstable angina (within 12 months of study entry)
  * New York Heart Association (NYHA) grade II or higher congestive heart failure
  * Evidence of bleeding diathesis/coagulopathy
  * Serious non-healing wound or bone fracture
* Patients with a history of the following within 28 days prior to registration are not eligible:

  * Abdominal fistula
  * Gastrointestinal perforation
  * Intrabdominal abscess
* Patients with a history of the following within 28 days prior to day 0 (first treatment day) are not eligible:

  * Major surgical procedure
  * Open biopsy
  * Significant traumatic injury
* Patients must not have core biopsy within 7 days prior to day 0 (first treatment day)
* Patients with prothrombin time (PT) (international normalized ratio [INR]) > 1.5 are not eligible, unless the patient is on full-dose anticoagulants; if so, the following criteria must be met for enrollment:

  * The subject must have an in-range INR (usually between 2 and 3), be on a stable dose of warfarin or on a stable dose of low molecular weight heparin
  * The subject must not have active bleeding or a pathological condition that is associated with a high risk of bleeding

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 57 (Actual)
Dates: Start 2006-07-25 (Actual); Primary Completion 2013-08-12 (Actual); Study Completion 2019-02-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jerome C Landry, Principal Investigator — ECOG-ACRIN Cancer Research Group
Locations (107):
- United States (107):
  - University of Alabama at Birmingham Cancer Center, Birmingham, Alabama
  - The Hospital of Central Connecticut, New Britain, Connecticut
  - Emory University Hospital/Winship Cancer Institute, Atlanta, Georgia
  - Atlanta VA Medical Center, Decatur, Georgia
  - Medical Center of Central Georgia, Macon, Georgia
  - Rush - Copley Medical Center, Aurora, Illinois
  - MacNeal Hospital and Cancer Center, Berwyn, Illinois
  - Hematology and Oncology Associates, Chicago, Illinois
  - Northwestern University, Chicago, Illinois
  - Jesse Brown Veterans Affairs Medical Center, Chicago, Illinois
  - Mercy Hospital and Medical Center, Chicago, Illinois
  - Swedish Covenant Hospital, Chicago, Illinois
  - Presence Saint Joseph Hospital-Chicago, Chicago, Illinois
  - Saint Anthony Memorial Hospital, Effingham, Illinois
  - Hematology Oncology Associates of Illinois-Highland Park, Highland Park, Illinois
  - Hinsdale Hematology Oncology Associates Incorporated, Hinsdale, Illinois
  - Midwest Center for Hematology Oncology, Joliet, Illinois
  - Joliet Oncology-Hematology Associates Limited, Joliet, Illinois
  - NorthShore Hematology Oncology-Libertyville, Libertyville, Illinois
  - Garneau, Stewart C MD (UIA Investigator), Moline, Illinois
  - Porubcin, Michael MD (UIA Investigator), Moline, Illinois
  - Sharis, Christine M MD (UIA Investigator), Moline, Illinois
  - Spector, David MD (UIA Investigator), Moline, Illinois
  - Stoffel, Thomas J MD (UIA Investigator), Moline, Illinois
  - Trinity Medical Center, Moline, Illinois
  - Vigliotti, Antonio, P.G. M.D. (UIA Investigator), Moline, Illinois
  - DuPage Medical Group-Ogden, Naperville, Illinois
  - Illinois Cancer Specialists-Niles, Niles, Illinois
  - Edward H Kaplan MD and Associates, Skokie, Illinois
  - Hematology Oncology Associates of Illinois - Skokie, Skokie, Illinois
  - Carle Cancer Center, Urbana, Illinois
  - Franciscan Saint Anthony Health-Michigan City, Michigan City, Indiana
  - Constantinou, Costas L MD (UIA Investigator), Bettendorf, Iowa
  - Siouxland Regional Cancer Center, Sioux City, Iowa
  - Mercy Medical Center-Sioux City, Sioux City, Iowa
  - Saint Luke's Regional Medical Center, Sioux City, Iowa
  - Bronson Methodist Hospital, Kalamazoo, Michigan
  - West Michigan Cancer Center, Kalamazoo, Michigan
  - Borgess Medical Center, Kalamazoo, Michigan
  - Fairview Ridges Hospital, Burnsville, Minnesota
  - Mercy Hospital, Coon Rapids, Minnesota
  - Fairview-Southdale Hospital, Edina, Minnesota
  - Unity Hospital, Fridley, Minnesota
  - Hutchinson Area Health Care, Hutchinson, Minnesota
  - Meeker County Memorial Hospital, Litchfield, Minnesota
  - Minnesota Oncology Hematology PA-Maplewood, Maplewood, Minnesota
  - Saint John's Hospital - Healtheast, Maplewood, Minnesota
  - Abbott-Northwestern Hospital, Minneapolis, Minnesota
  - Virginia Piper Cancer Institute, Minneapolis, Minnesota
  - Hennepin County Medical Center, Minneapolis, Minnesota
  - North Memorial Medical Health Center, Robbinsdale, Minnesota
  - Metro Minnesota Community Oncology Research Consortium, Saint Louis Park, Minnesota
  - Park Nicollet Clinic - Saint Louis Park, Saint Louis Park, Minnesota
  - Regions Hospital, Saint Paul, Minnesota
  - Saint Joseph's Hospital - Healtheast, Saint Paul, Minnesota
  - United Hospital, Saint Paul, Minnesota
  - Saint Francis Regional Medical Center, Shakopee, Minnesota
  - Ridgeview Medical Center, Waconia, Minnesota
  - Minnesota Oncology Hematology PA-Woodbury, Woodbury, Minnesota
  - Woodwinds Health Campus, Woodbury, Minnesota
  - Nebraska Cancer Research Center, Lincoln, Nebraska
  - Missouri Valley Cancer Consortium, Omaha, Nebraska
  - Alegent Health Immanuel Medical Center, Omaha, Nebraska
  - Alegent Health Bergan Mercy Medical Center, Omaha, Nebraska
  - Creighton University Medical Center, Omaha, Nebraska
  - Virtua Memorial, Mount Holly, New Jersey
  - Sparta Cancer Treatment Center, Sparta, New Jersey
  - Virtua Voorhees, Voorhees Township, New Jersey
  - Inspira Medical Center Woodbury, Woodbury, New Jersey
  - Montefiore Medical Center-Wakefield Campus, The Bronx, New York
  - Montefiore Medical Center - Moses Campus, The Bronx, New York
  - Summa Akron City Hospital/Cooper Cancer Center, Akron, Ohio
  - Summa Barberton Hospital, Barberton, Ohio
  - Mary Rutan Hospital, Bellefontaine, Ohio
  - Adena Regional Medical Center, Chillicothe, Ohio
  - Riverside Methodist Hospital, Columbus, Ohio
  - Grant Medical Center, Columbus, Ohio
  - Mount Carmel Health Center West, Columbus, Ohio
  - Doctors Hospital, Columbus, Ohio
  - Grady Memorial Hospital, Delaware, Ohio
  - Fairfield Medical Center, Lancaster, Ohio
  - Saint Rita's Medical Center, Lima, Ohio
  - Marietta Memorial Hospital, Marietta, Ohio
  - Licking Memorial Hospital, Newark, Ohio
  - Springfield Regional Medical Center, Springfield, Ohio
  - Saint Ann's Hospital, Westerville, Ohio
  - Genesis Healthcare System Cancer Care Center, Zanesville, Ohio
  - Natalie Warren Bryant Cancer Center at Saint Francis, Tulsa, Oklahoma
  - Lehigh Valley Hospital-Cedar Crest, Allentown, Pennsylvania
  - Mercy Fitzgerald Hospital, Darby, Pennsylvania
  - Pocono Medical Center, East Stroudsburg, Pennsylvania
  - Ephrata Cancer Center, Ephrata, Pennsylvania
  - Riddle Memorial Hospital, Media, Pennsylvania
  - Thomas Jefferson University Hospital, Philadelphia, Pennsylvania
  - Fox Chase Cancer Center, Philadelphia, Pennsylvania
  - Aria Health-Torresdale Campus, Philadelphia, Pennsylvania
  - Einstein Medical Center Philadelphia, Philadelphia, Pennsylvania
  - Hematology and Oncology Associates of North East Pennsylvania, Scranton, Pennsylvania
  - Associates In Hematology Oncology PC-Upland, Upland, Pennsylvania
  - Sanford Cancer Center Oncology Clinic, Sioux Falls, South Dakota
  - Avera Cancer Institute, Sioux Falls, South Dakota
  - Avera McKennan Hospital and University Health Center, Sioux Falls, South Dakota
  - Medical X-Ray Center, Sioux Falls, South Dakota
  - Sanford USD Medical Center - Sioux Falls, Sioux Falls, South Dakota
  - UT Southwestern/Simmons Cancer Center-Dallas, Dallas, Texas
  - Gundersen Lutheran Medical Center, La Crosse, Wisconsin
  - Froedtert and the Medical College of Wisconsin, Milwaukee, Wisconsin

REFERENCES:
- [Derived] Landry JC, Feng Y, Prabhu RS, Cohen SJ, Staley CA, Whittington R, Sigurdson ER, Nimeiri H, Verma U, Benson AB. Phase II Trial of Preoperative Radiation With Concurrent Capecitabine, Oxaliplatin, and Bevacizumab Followed by Surgery and Postoperative 5-Fluorouracil, Leucovorin, Oxaliplatin (FOLFOX), and Bevacizumab in Patients With Locally Advanced Rectal Cancer: 5-Year Clinical Outcomes ECOG-ACRIN Cancer Research Group E3204. Oncologist. 2015 Jun;20(6):615-6. doi: 10.1634/theoncologist.2015-0106. Epub 2015 Apr 29. PMID 25926352

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This study was activated on July 25, 2006 and terminated on May 26, 2010 with a final accrual of 57 patients from 11 participating sites.
Groups:
- Arm I: Preoperative radiation therapy: Patients undergo radiotherapy once daily 5 days a week.
  Preoperative chemotherapy: Patients receive oral capecitabine twice daily 5 days a week for 5.5 weeks. Patients also receive oxaliplatin IV over 2 hours on days 1, 8, 15, 22, and 29 and bevacizumab IV over 30-90 minutes on days 1, 15, and 29 during radiotherapy.
  Surgery: Approximately 6-8 weeks after completion of chemoradiotherapy, patients undergo surgical resection.
  Postoperative chemotherapy: Approximately 4-12 weeks after surgery, patients receive oxaliplatin IV over 2 hours, leucovorin calcium IV over 2 hours, bevacizumab IV over 30-90 minutes on day 1. Patients also receive fluorouracil (5-FU) IV continuously over 46 hours beginning on day 1. Treatment repeats every 2 weeks for 9 courses. Patients then receive up to 3 additional courses of leucovorin calcium, 5-FU, and bevacizumab.
  radiation therapy: Patients undergo 3-dimensional conformal radiation therapy once daily 5 days
Period: Overall Study
Arm/Group | Arm I
Started | 57
Eligible | 55
Started Protocol Therapy | 55
Eligible and Treated | 53
Completed | 18
Not Completed | 39
Not completed — Adverse Event | 18
Not completed — Death | 2
Not completed — Withdrawal by Subject | 8
Not completed — Alternative therapy | 1
Not completed — Complicating disese | 1
Not completed — Other | 5
Not completed — Not start protocol therapy | 2
Not completed — Ineligible | 2

BASELINE CHARACTERISTICS:
Population: Eligible and treated patients
Groups:
- Arm I: Preoperative radiation therapy: Patients undergo radiotherapy once daily 5 days a week.
  Preoperative chemotherapy: Patients receive oral capecitabine twice daily 5 days a week for 5.5 weeks. Patients also receive oxaliplatin IV over 2 hours on days 1, 8, 15, 22, and 29 and bevacizumab IV over 30-90 minutes on days 1, 15, and 29 during radiotherapy.
  Surgery: Approximately 6-8 weeks after completion of chemoradiotherapy, patients undergo surgical resection.
  Postoperative chemotherapy: Approximately 4-8 weeks after surgery, patients receive oxaliplatin IV over 2 hours, leucovorin calcium IV over 2 hours, and bevacizumab IV over 30-90 minutes on day 1. Patients also receive fluorouracil (5-FU) IV continuously over 46 hours beginning on day 1. Treatment repeats every 2 weeks for 9 courses. Patients then receive up to 3 additional courses of leucovorin calcium, 5-FU, and bevacizumab.
Arm/Group | Arm I
Number analyzed (Participants) | 53
Age, Continuous [Median (Full Range); unit: years] | 54 [25 to 83]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 17
  Male | 36
Clinical T stage [Number; unit: participants]
  T3 | 49
  T4 | 4

OUTCOME MEASURES:

1. Primary Outcome: Pathologic Complete Response Rate
Description: Pathologic complete response to preoperative therapy was determined at the time of surgical resection. Pathologic complete response (pCR) is defined as no evidence of invasive cells on pathologic examination of the primary rectal cancer (or tissue from the area where the tumor had been if there is a complete clinical response). Pathologic complete response rate is calculated as number of patients achieving pathologic complete response divided by all eligible and treated patients
Time Frame: Assessed at surgery time
Population: Eligible and treated patients
Measure: Number (90% Confidence Interval); unit: percentage of participants
Groups:
- Arm I: Preoperative radiation therapy: Patients undergo radiotherapy once daily 5 days a week.
  Preoperative chemotherapy: Patients receive oral capecitabine twice daily 5 days a week for 5.5 weeks. Patients also receive oxaliplatin IV over 2 hours on days 1, 8, 15, 22, and 29 and bevacizumab IV over 30-90 minutes on days 1, 15, and 29 during radiotherapy.
  Surgery: Approximately 6-8 weeks after completion of chemoradiotherapy, patients undergo surgical resection.
  Postoperative chemotherapy: Approximately 4-12 weeks after surgery, patients receive oxaliplatin IV over 2 hours, leucovorin calcium IV over 2 hours, and bevacizumab IV over 30-90 minutes on day 1. Patients also receive fluorouracil (5-FU) IV continuously over 46 hours beginning on day 1. Treatment repeats every 2 weeks for 9 courses. Patients then receive up to 3 additional courses of leucovorin calcium, 5-FU, and bevacizumab.
Arm/Group | Arm I
Number analyzed (Participants) | 53
percentage of participants | 17 [7 to 32]

2. Secondary Outcome: Resection Rate for T3 Rectal Cancers
Description: Resection rate is defined as number of patients with T3 rectal cancer who underwent curative surgical resection among all eligible and treated patients with T3 rectal cancers
Time Frame: Assessed at surgery time
Population: eligible and treated patients with T3 rectal cancers
Measure: Number (90% Confidence Interval); unit: percentage of participants
Arm/Group | Arm I
Number analyzed (Participants) | 49
percentage of participants | 92 [82 to 97]

3. Secondary Outcome: Resection Rate for T4 Rectal Cancers
Description: Resection rate is defined as number of patients with T4 rectal cancer who underwent curative surgical resection among all eligible and treated patients with T4 rectal cancers
Time Frame: Assessed at surgery time
Population: eligible and treated patients with T4 rectal cancers
Measure: Number (90% Confidence Interval); unit: percentage of participants
Arm/Group | Arm I
Number analyzed (Participants) | 4
percentage of participants | 75 [25 to 99]

4. Secondary Outcome: 5-year Overall Survival Rate
Description: Overall survival is defined as time from registration to death from any cause. 5-year overall survival rate is estimated using Kaplan-Meier method.
Time Frame: survival follow-up began after post-operative chemotherapy, assessed every 3 months for patients 3-5 years from registration, every 6 months for patients 5-10 years from registration and every 12 months for patients 10 years from registration
Population: Eligible and treated patients
Measure: Number (90% Confidence Interval); unit: percentage of participants
Arm/Group | Arm I
Number analyzed (Participants) | 53
percentage of participants | 80 [67 to 92]

5. Secondary Outcome: 5-year Recurrence-free Survival Rate
Description: Recurrence free survival is defined as time from surgery to disease recurrence or death without recurrence (whichever occurred first) among resected patients. 5-year recurrence-free survival rate is estimated using Kaplan-Meier method, with 90% confidence interval calculated using Greenwood's formula.
Time Frame: recurrence follow-up began after post-operative chemotherapy, assessed every 3 months for patients 3-5 years from registration, every 6 months for patients 5-10 years from registration and every 12 months for patients 10 years from registration
Population: Eligible and treated patients who underwent surgery after neoadjuvant therapy
Measure: Number (90% Confidence Interval); unit: percentage of participants
Arm/Group | Arm I
Number analyzed (Participants) | 48
percentage of participants | 81 [68 to 94]

ADVERSE EVENTS:
Time Frame: Assessed at the completion of Pre-Operative Chemoradiation, at the end of every cycle during PostOperative Chemotherapy, and at 30 days after the end of treatment
Description: Prior to diagnosis of progression/relapse, any severe (Grade ≥ 3) long term toxicity that has not been previously reported were collected using the Long-term follow up form.
Arm/Group | Arm I
Serious Adverse Events (participants affected / at risk) | 39/55
Other Adverse Events (participants affected / at risk) | 53/55
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Arm I (N=55)
Allergic reaction (Immune system disorders) | 1
Anemia (Blood and lymphatic system disorders) | 5
Leukocytes decreased (Investigations) | 8
Lymphopenia (Investigations) | 8
Neutrophils decreased (Investigations) | 10
Platelets decreased (Investigations) | 3
Fatigue (General disorders) | 9
Hypothermia (General disorders) | 1
Weight loss (Investigations) | 2
DIC (Blood and lymphatic system disorders) | 1
Coagulation-other (Investigations) | 1
Rash/desquamation (Skin and subcutaneous tissue disorders) | 2
Chemoradiation dermatitis (Injury, poisoning and procedural complications) | 1
Wound - non-infectious (Injury, poisoning and procedural complications) | 2
Skin-other (Skin and subcutaneous tissue disorders) | 1
Death NOS (General disorders) | 1
Anorexia (Metabolism and nutrition disorders) | 2
Constipation (Gastrointestinal disorders) | 1
Dehydration (Metabolism and nutrition disorders) | 5
Diarrhea w/o prior colostomy (Gastrointestinal disorders) | 7
Distention/bloating, abdominal (Gastrointestinal disorders) | 1
Enteritis (Gastrointestinal disorders) | 1
Fistula, Rectum (Gastrointestinal disorders) | 1
Ileus (Gastrointestinal disorders) | 2
Nausea (Gastrointestinal disorders) | 3
Proctitis (Gastrointestinal disorders) | 1
Vomiting (Gastrointestinal disorders) | 3
CNS, hemorrhage (Nervous system disorders) | 1
Oral cavity, hemorrhage (Gastrointestinal disorders) | 1
Infection Gr0-2 neut, anal/perianl (Infections and infestations) | 1
Infection Gr0-2 neut, muscle (Infections and infestations) | 1
Infection Gr0-2 neut, pelvis NOS (Infections and infestations) | 1
Infection Gr0-2 neut, rectum (Infections and infestations) | 1
Infection Gr0-2 neut, wound (Infections and infestations) | 2
Infection w/ unk ANC anal/perianal (Infections and infestations) | 2
Infection w/ unk ANC wound (Infections and infestations) | 1
Acidosis (Metabolism and nutrition disorders) | 1
Hypoalbuminemia (Metabolism and nutrition disorders) | 2
Alkaline phosphatase increased (Investigations) | 1
Aspartate aminotransferase increased (Investigations) | 1
Hypocalcemia (Metabolism and nutrition disorders) | 1
Hyperglycemia (Metabolism and nutrition disorders) | 2
Hypophosphatemia (Metabolism and nutrition disorders) | 1
Hyperkalemia (Metabolism and nutrition disorders) | 2
Hyponatremia (Metabolism and nutrition disorders) | 1
Metabolic/Laboratory-other (Investigations) | 1
Neuropathy-motor (Nervous system disorders) | 1
Neuropathy-sensory (Nervous system disorders) | 5
Abdomen, pain (Gastrointestinal disorders) | 5
Bone, pain (Musculoskeletal and connective tissue disorders) | 1
Intestine, pain (Gastrointestinal disorders) | 1
Perineum, pain (Reproductive system and breast disorders) | 1
Rectum, pain (Gastrointestinal disorders) | 9
Pain-other (General disorders) | 1
Aspiration (Respiratory, thoracic and mediastinal disorders) | 1
Incontinence urinary (Renal and urinary disorders) | 1
Renal failure (Renal and urinary disorders) | 1
Urinary retention (Renal and urinary disorders) | 1
Erectile impotence (Reproductive system and breast disorders) | 1
Thrombosis/thrombus/embolism (Vascular disorders) | 2
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Arm I (N=55)
Anemia (Blood and lymphatic system disorders) | 33
Leukocytes decreased (Investigations) | 23
Lymphopenia (Investigations) | 7
Neutrophils decreased (Investigations) | 17
Platelets decreased (Investigations) | 22
Hypotension (Vascular disorders) | 4
Fatigue (General disorders) | 31
Fever w/o neutropenia (General disorders) | 5
Insomnia (Psychiatric disorders) | 5
Rigors/chills (General disorders) | 3
Sweating (Skin and subcutaneous tissue disorders) | 4
Weight loss (Investigations) | 17
Dry skin (Skin and subcutaneous tissue disorders) | 3
Alopecia (Skin and subcutaneous tissue disorders) | 4
Hyperpigmentation (Skin and subcutaneous tissue disorders) | 3
Rash/desquamation (Skin and subcutaneous tissue disorders) | 7
Hand-foot reaction (Skin and subcutaneous tissue disorders) | 3
Wound - non-infectious (Injury, poisoning and procedural complications) | 6
Anorexia (Metabolism and nutrition disorders) | 17
Constipation (Gastrointestinal disorders) | 9
Dehydration (Metabolism and nutrition disorders) | 5
Diarrhea w/o prior colostomy (Gastrointestinal disorders) | 27
Dry mouth (Gastrointestinal disorders) | 3
Dyspepsia (Gastrointestinal disorders) | 5
Incontinence, anal (Gastrointestinal disorders) | 3
Muco/stomatitis (symptom) oral cavity (Gastrointestinal disorders) | 7
Nausea (Gastrointestinal disorders) | 23
Proctitis (Gastrointestinal disorders) | 5
Taste disturbance (Nervous system disorders) | 4
Vomiting (Gastrointestinal disorders) | 13
Rectum, hemorrhage (Gastrointestinal disorders) | 4
Urinary hemorrhage NOS (Renal and urinary disorders) | 3
Nose, hemorrhage (Respiratory, thoracic and mediastinal disorders) | 3
Hypoalbuminemia (Metabolism and nutrition disorders) | 4
Alkaline phosphatase increased (Investigations) | 3
Alanine aminotransferase increased (Investigations) | 5
Aspartate aminotransferase increased (Investigations) | 11
Hypocalcemia (Metabolism and nutrition disorders) | 7
Hyperglycemia (Metabolism and nutrition disorders) | 5
Hypokalemia (Metabolism and nutrition disorders) | 6
Hyponatremia (Metabolism and nutrition disorders) | 4
Metabolic/Laboratory-other (Investigations) | 3
Dizziness (Nervous system disorders) | 3
Depression (Psychiatric disorders) | 3
Neuropathy-sensory (Nervous system disorders) | 28
Abdomen, pain (Gastrointestinal disorders) | 9
Back, pain (Musculoskeletal and connective tissue disorders) | 3
Head/headache (Nervous system disorders) | 5
Rectum, pain (Gastrointestinal disorders) | 14
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 5
Voice changes/dysarthria (Respiratory, thoracic and mediastinal disorders) | 3
Urinary frequency/urgency (Renal and urinary disorders) | 6

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less